CLINICAL TRIAL: NCT05534204
Title: Evaluation of the Effects of Silk and Polyester Suture on Postoperative Complications in Lower Impacted Third Molar Surgery
Brief Title: Evaluation of the Effects of Silk and Polyester Suture on Postoperative Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, levent Cigerim, Head of Oral and Maxillofacial Surgery Department, Yuzuncu Yil University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 21.05.2020/06
Record Dates: First submitted 2022-02-14; First posted 2022-09-09 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silk suture (Active Comparator): Silk suture is a multifilament suture, used for surgical sides closure.
  Interventions: Procedure: Silk suture
- Polyester suture (Active Comparator): Polyester suture is a monofilament suture, used for surgical sides closure.
  Interventions: Procedure: Polyester suture

INTERVENTIONS:
Procedure: Silk suture — Patients with bilateral impacted lower third molars will have operations for both sides. On one side for primarily closure after operation silk suture will be used.
  Arms: Silk suture
Procedure: Polyester suture — Patients with bilateral impacted lower third molars will have operations for both side. On one side for primarily closure after operation polyester suture will be used.
  Arms: Polyester suture

SUMMARY:
Some undesirable complications such as pain, swelling, trismus, paresthesia, hematoma, infection and, albeit rare, fractures may occur after lower impacted wisdom tooth surgery. More effective wound closure methods with fewer complications have positive effects on postoperative recovery. Suturing is the most commonly used wound closure technique after lower impacted wisdom tooth surgery. Suturing, which is the last step of the operation, contributes to wound healing in order to reposition and stabilize the tissue components and to control bleeding. In our study, it was aimed to evaluate the efficacy of silk and polyester sutures used in wound closure techniques, which are frequently used in lower impacted wisdom teeth surgery.

DETAILED DESCRIPTION:
This randomized, single-blind, split-mouth study was carried out on 30 patients who applied to Van Yuzuncu Yıl University, Faculty of Dentistry, Department of Oral, Dental and Maxillofacial Surgery. Silk suture was used on one side of the patients and polyester suture was used on the other side. When the patients first applied to the clinic, their anamnesis was taken and panoramic images were taken after clinical evaluations were made.

Evaluations were made with preoperative face measurements (for evaluation of swelling), maximum mouth opening (for evaluation of trismus) and periodontal measurements for all patients. The mentioned measurements and evaluations were repeated on the 2nd and 7th postoperative days. In addition, postoperative pain was evaluated with the VAS scale.

The same surgical procedure was performed by the same surgeon for all patients. After local anesthesia (2ml of 80 mg Articaine hydrochloride + 0.02mg Epinephrine bitartrate) a 3-corner flap containing the vertical incision passing through the mesial of the number 7 was lifted, the bone removed under saline cooling and the teeth were separated when needed. Afterwards, the extraction sockets will be irrigated with saline to control bleeding, and the area is closed primarily with silk or polyester suture material.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and over
* Impacted teeth in mesial and horizontal positions and in class 2 and class B according to Pell & Gregory classification,
* Asymptomatic impacted teeth,
* Individuals who is coming to control and fill in the given and requested forms,
* Individuals with an operation time of 30 minutes or less

Exclusion Criteria:

* Systemic disease,
* Smoking,
* Pregnancy or breastfeeding,
* Allergy to the drugs to be used in the study,
* Using any additional medication that may affect the outcome of the study,
* Using medication until 2 weeks before the operations,
* Post-operative alveolitis.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Postoperative1st day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperative 2nd day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperative 3rd day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperative 5th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperative 7th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analogue scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Levent Ciğerim, Assoc.Prof., Principal Investigator — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University, Faculty of Dentistry, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT05534204/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT05534204/ICF_001.pdf